CLINICAL TRIAL: NCT03800173
Title: A Phase 1 Double-blind, Placebo Controlled, Dose Ranging Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Galidesivir (BCX4430) Administered as Single Doses Via Intravenous Infusion in Healthy Subjects
Brief Title: A Study to Evaluate the Single Dose Safety, Tolerability and Pharmacokinetics of IV BCX4430
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCX4430-106; DMID18-0013 (Other: NIAID); 272201300017C-18-0-1 (NIH)
Record Dates: First submitted 2018-12-12; First posted 2019-01-11 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Marburg Virus Disease
MeSH Terms: conditions — Marburg Virus Disease | interventions — galidesivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Galidesivir (Experimental): Galidesivir IV infusion
  Interventions: Drug: galidesivir
- placebo (Placebo Comparator): Placebo IV infusion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: galidesivir — galidesivir IV infusion
  Arms: Galidesivir
Drug: placebo — placebo IV infusion
  Arms: placebo

SUMMARY:
This is a placebo-controlled, randomized, double-blind study to evaluate the pharmacokinetics of galidesivir following administration of single doses by IV infusion

DETAILED DESCRIPTION:
This single ascending dose study will evaluate the safety, tolerability, and PK of single doses of galidesivir vs. placebo administered as IV infusions in healthy subjects enrolled in up to four dose cohorts of 8 subjects each. A single dose of study drug will be administered per cohort: 6 subjects will receive galidesivir IV, and 2 subjects will receive matching placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* written informed consent
* males and non-pregnant, non-lactating females
* BMI 19.0-32.0
* willing to abide by contraceptive requirements
* normal vitals
* willing to abide by study procedures and restrictions

Exclusion Criteria:

* clinically significant medical condition or medical history or psychiatric condition or history of psychiatric condition
* abnormal cardiac finding, or laboratory/urinalysis abnormality at screening
* known family history of sudden death or long QT syndrome, family or personal history of QT prolongation, or arrhythmia that required medical intervention
* current participation in any other investigational drug study or participation in an investigational drug study within 3 months of screening visit
* use of prescription, OTC, or herbal medications during study or use of any specified medications within 30 days prior to study
* Recent or current history of alcohol or drug abuse
* Regular use of tobacco or nicotine products
* Positive serology for HBV, HCV, or HIV
* history of severe adverse reaction to or known sensitivity to any drug
* pregnant, lactating, or planning to become pregnant within 30 days of the study. Male subjects with pregnant female partners are excluded

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dickerson, MD, PhD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mathis A, Collins D, Dobo S, Walling DM, Sheridan WP, Taylor R. Pharmacokinetics and Safety of the Nucleoside Analog Antiviral Drug Galidesivir Administered to Healthy Adult Subjects. Clin Pharmacol Drug Dev. 2022 Apr;11(4):467-474. doi: 10.1002/cpdd.1037. Epub 2022 Feb 19. PMID 35182042

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A single dose of study drug was administered to subjects in each of cohorts 1 to 4. In each cohort, 6 subjects received galidesivir and 2 subjects received matching placebo.
Groups:
- Placebo: single placebo IV infusion
- 5 mg/kg Galidesivir: Single IV infusion 5 mg/kg galidesivir
- 10 mg/kg Galidesivir: Single IV infusion 10 mg/kg galidesivir
- 15 mg/kg Galidesivir: Single IV infusion 15 mg/kg galidesivir
- 20 mg/kg Galidesivir: Single IV infusion 20 mg/kg galidesivir
Period: Overall Study
Arm/Group | Placebo | 5 mg/kg Galidesivir | 10 mg/kg Galidesivir | 15 mg/kg Galidesivir | 20 mg/kg Galidesivir
Started | 8 | 6 | 6 | 6 | 6
Safety Population (Safety Population includes all subjects who received study drug.) | 8 | 6 | 6 | 6 | 6
PK Population (PK population included all subjects from whom at least 1 galidesivir PK parameter was estimated.) | 0 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized subjects who received any amount of study drug (i.e. a partial infusion). Subjects were analyzed according to the treatment received. The safety population was used for analyses of demographics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 mg/kg Galidesivir | 10 mg/kg Galidesivir | 15 mg/kg Galidesivir | 20 mg/kg Galidesivir | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (6.88) | 39.8 (10.76) | 33.5 (8.76) | 41.7 (12.04) | 31.8 (8.98) | 35.3 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 1 | 2 | 2 | 13
  Male | 3 | 3 | 5 | 4 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 3 | 0 | 3 | 12
  White | 2 | 5 | 3 | 6 | 3 | 19
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Galidesivir Safety and Tolerability, as Measured by the Number of Participants Experiencing Adverse Events.
Description: Any event reported on the subject's study record that occurred on or after the initiation of study drug was defined as treatment emergent (TEAE).
Time Frame: AEs were assessed and recorded from the time of signing the ICF through to the appropriate follow-up period, up to 23 days from IMP dosing on Day 1.
Population: The safety population included all randomized subjects who received any amount of study drug (i.e. a partial infusion).
Measure: Number; unit: participants
Arm/Group | Placebo | 5 mg/kg Galidesivir | 10 mg/kg Galidesivir | 15 mg/kg Galidesivir | 20 mg/kg Galidesivir
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
participants
  Subjects with at least 1 TEAE | 2 | 0 | 1 | 4 | 1
  Not related TEAEs | 2 | 0 | 1 | 2 | 0
  Related TEAEs | 0 | 0 | 0 | 2 | 1
  Mild TEAE | 2 | 0 | 1 | 3 | 1
  Moderate TEAE | 0 | 0 | 0 | 0 | 0
  Severe TEAE | 0 | 0 | 0 | 1 | 0
  Subjects with at least 1 SAE | 0 | 0 | 1 | 1 | 0
  Subject Discontinuation due to AE | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Plasma PK - Galidesivir Cmax (Maximum Observed Concentration of Drug)
Description: Serial blood samples for PK assessment of plasma galidesivir were collected at the following time points:
  * Day 1 to Day 5: 0 hour (pre dose), halfway through the infusion (0.5 hour), 1 hour (end of the infusion), 1.25, 1.50, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 60, 72, and 96 hours post dose.
  * Day 6 (+1 day), Day 8 (+1 day), Day 14 (± 1 day)
  * Day 21 (+2 days) or early termination.
  Cmax for galidesivir was estimated using non compartmental methods with Phoenix® WinNonlin® v8.1 or higher (Certara, Inc.).
Time Frame: Plasma PK parameters are based on sampling over a 21 day period
Population: The PK population included subjects for whom at least 1 PK parameter was estimated. The PK population was the primary population for the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 5 mg/kg Galidesivir | 10 mg/kg Galidesivir | 15 mg/kg Galidesivir | 20 mg/kg Galidesivir
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 5540 (7.8) | 10300 (22.3) | 17730 (17.5) | 20490 (16.2)
Statistical Analysis 1: Comparison: 5 mg/kg Galidesivir vs 10 mg/kg Galidesivir vs 15 mg/kg Galidesivir vs 20 mg/kg Galidesivir; A model with In-transformed dose (dose continuous) as a fixed effect & subject as a random effect was applied to In-transformed Cmax. Dose proportionality was assessed by restricted max likelihood using SAS PROC MIXED. The mean slope was estimated from the power model & the corresponding 90% CI calculated. Although there was no formal statistical hypothesis tested for this secondary objective, there was evidence for dose proportionality if the 90% CI of the fixed slope for In-dose contained 1; Test type: Other; Slope = 0.982, 90% CI 2-sided [0.868 to 1.096]

3. Secondary Outcome: Plasma PK - Galidesivir AUC (Area Under the Concentration vs. Time Curve)
Description: Serial blood samples for PK assessment of plasma galidesivir were collected at the following time points:
  * Day 1 to Day 5: 0 hour (pre dose), halfway through the infusion (0.5 hour), 1 hour (end of the infusion), 1.25, 1.50, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 60, 72, and 96 hours post dose.
  * Day 6 (+1 day), Day 8 (+1 day), Day 14 (± 1 day)
  * Day 21 (+2 days) or early termination.
  AUC0-inf (AUC from time 0 extrapolated to infinite time) and AUC0-t (AUC from time 0 to time t, where "t" = the last quantifiable concentration) for galidesivir was estimated using non compartmental methods with Phoenix® WinNonlin® v8.1 or higher (Certara, Inc.).
Time Frame: Plasma PK parameters are based on sampling over a 21 day period
Population: The PK population included subjects for whom at least 1 PK parameter was estimated. The PK population was the primary population for the PK analysis. Only 5 subjects were included in the 20 mg/kg cohort for AUC0-t analysis, as 1 subject was lost to follow-up after discharge from clinic on Day 5.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 5 mg/kg Galidesivir | 10 mg/kg Galidesivir | 15 mg/kg Galidesivir | 20 mg/kg Galidesivir
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*h/mL
  AUC0-inf | 21160 (23.0) | 37080 (14.5) | 65860 (21.9) | 81230 (14.3)
  AUC0-t: number analyzed (Participants) | 6 | 6 | 6 | 5
  AUC0-t | 17150 (21.0) | 32360 (17.4) | 59590 (22.0) | 73350 (14.1)
Statistical Analysis 1: Comparison: 5 mg/kg Galidesivir vs 10 mg/kg Galidesivir vs 15 mg/kg Galidesivir vs 20 mg/kg Galidesivir; A model with In-transformed dose (dose continuous) as a fixed effect & subject as a random effect was applied to In-transformed AUC0-inf Dose proportionality was assessed by restricted max likelihood using SAS PROC MIXED. The mean slope was estimated from the power model & the corresponding 90% CI calculated. Although there was no formal statistical hypothesis tested for this secondary objective, there was evidence for dose proportionality if the 90% CI of the fixed slope for In-dose contained 1; Test type: Other; Slope = 1.000, 90% CI 2-sided [0.872 to 1.128]
Statistical Analysis 2: Comparison: 5 mg/kg Galidesivir vs 10 mg/kg Galidesivir vs 15 mg/kg Galidesivir vs 20 mg/kg Galidesivir; A model with In-transformed dose (dose continuous) as a fixed effect & subject as a random effect was applied to In-transformed AUC0-t. Dose proportionality was assessed by restricted max likelihood using SAS PROC MIXED. The mean slope was estimated from the power model & the corresponding 90% CI calculated. Although there was no formal statistical hypothesis tested for this secondary objective, there was evidence for dose proportionality if the 90% CI of the fixed slope for In-dose contained 1; Test type: Other; Slope = 1.086, 90% CI 2-sided [0.952 to 1.219]

4. Secondary Outcome: Galidesivir Renal Clearance
Description: Urine was collected from subjects over a 96 hour period per protocol, analyzed for galidesivir concentrations. Urine PK parameters including CLR (renal clearance of unchanged drug cumulatively over all collection intervals or in a specific interval) were estimated in SAS for Windows v9.4 or higher (SAS Institute, Inc.) based on the recorded urine concentrations and volumes.
Time Frame: Urine PK parameters are based on sampling over a 96 hour period.
Population: The PK population included subjects for whom at least 1 PK parameter was estimated. The PK population was the primary population for the PK analysis. There were only 5 subjects in the 20 mg/kg cohort as 1 subject was lost to follow-up after discharge from clinic on Day 5.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | 5 mg/kg Galidesivir | 10 mg/kg Galidesivir | 15 mg/kg Galidesivir | 20 mg/kg Galidesivir
Number analyzed (Participants) | 6 | 6 | 6 | 5
L/hr | 9.305 (16.7) | 11.66 (17.8) | 11.51 (14.5) | 7.131 (90.4)

ADVERSE EVENTS:
Time Frame: AEs were assessed and recorded from the time of signing the ICF through to the appropriate follow-up visit, up to 23 days from IMP dosing on Day 1. All AEs were graded for severity using the modified 2014 DMID Adult Toxicity Grading Scale. Any AEs not covered by the DMID criteria were assessed and classified into 1 of 3 clearly defined categories (mild, moderate, or severe).
Arm/Group | Placebo | 5 mg/kg Galidesivir | 10 mg/kg Galidesivir | 15 mg/kg Galidesivir | 20 mg/kg Galidesivir
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 1/6 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/8 | 0/6 | 0/6 | 4/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 5 mg/kg Galidesivir (N=6) | 10 mg/kg Galidesivir (N=6) | 15 mg/kg Galidesivir (N=6) | 20 mg/kg Galidesivir (N=6)
gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 5 mg/kg Galidesivir (N=6) | 10 mg/kg Galidesivir (N=6) | 15 mg/kg Galidesivir (N=6) | 20 mg/kg Galidesivir (N=6)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03800173/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03800173/SAP_001.pdf